CLINICAL TRIAL: NCT03466723
Title: Novel and Minimal Invasive Biomarkers for Parkinson's Disease: Profiling of Serum Circulating miRNAs and Patho-physiological Implications
Brief Title: miRNAs Profiling in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Daniela Ruggiero, Ph.D., Neuromed IRCCS
Other Study IDs: DRPAR01
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — DNA, RNA, Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: biomarker identification in Parkinson disease — circulating miRNAs profiling by NGS analysis functional miRNA characterization association of miRNA levels with genetic variants

SUMMARY:
microRNAs (miRNAs) regulate fundamental cell processes. Dysregulation of miRNA expression and function is reported in various diseases including cancer, metabolic disorders as well as neurological disorders. Circulating miRNAs have been proposed to mirror physiological and pathological conditions suggesting their use as biomarkers for various diseases. The study will focus on a case-control study cohort (N=1000) of subjects recruited at the IRCCS Neuromed for which a deep clinical characterization and genome-wide sequencing data are available. This study will enable to identify novel circulating biomarkers for Parkinson's disease (PD). Further, the project will give new insights on the involvement of miRNAs in the etiology of PD and in the understanding of the genetics of the disease thus opening avenues for novel therapeutic strategies.

DETAILED DESCRIPTION:
Hypothesis and Significance:

The project intends to identify novel biomarkers for PD and clinical parameters related to the PD etiology. To do that circulating miRNA profiling through a next-generation sequencing will be performed using a single sample approach in the case-control study cohort and identified miRNAs will be validated by qRT-PCR and functional analyses. In addition, the project will contribute expanding the knowledge of the genetic architecture of PD taking advantage of genetic characterization of the study sample. miRNA genes and target genes will be used to prioritize genetic variants to be tested for association with PD to detect novel genes and functional variants that confer disease risk.

Specific Aim 1:

Profile of circulating miRNAs in the serum of PD patients and controls by next-generation sequencing in individual samples. Correlation between identified miRNAs and PD-related parameters and validation in independent cohorts

Specific Aim 2:

Bioinformatics prediction of target genes and miRNA functional validation

Specific Aim 3:

Identification of genes/genetic variants in miRNA pathways predisposing to PD

Expected outcomes:

The study will allow to discover novel circulating miRNAs as biomarkers for Parkinson's disease. As the deep phenotype characterization of the study sample, the project expects to find new associations of identified miRNAs with disease-related parameters and define the role of miRNAs in the physiological pathways in which those parameters are involved and in the etiology of PD. Also, the understanding of the genetics of the disease will open avenues for novel therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria for cases:

* Presence of at least two out the following cardinal signs: resting tremor, cogwheel rigidity, bradykinesia, asymmetrical onset of symptoms and symptomatic response to L-dopa (levodopa)

Exclusion Criteria for cases:

* Previous thalamotomy on the implanted sided, significant brain atrophy or structural damage seen on CT or MRI, marked cognitive dysfunction, active psychiatric symptoms, or concurrent neurological or other uncontrolled medical disorders.

Exclusion Criteria for controls:

Personal or family history for neurodegenerative diseases

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Collection of 1000 case-control study samples with a large phenotype and genotype characterization. The study includes 500 PD patients and 500 age/gender-matched controls. All PD patients have been diagnosed at the IRCCS Neuromed and followed-up (at least for 5 years) for disease progression. Data collected from patients and unrelated controls include: socio-demographic status, life style, anamnesis and family history, exposure to toxic chemical and/or environmental agents. Patients have been studied with a protocol comprising neurological examination (Stadio di Hoehn and Yahr, MDS-UPDRS part III, MOCA test) and evaluation of no motor symptoms. Information about drugs therapy have been also collected.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Identification of novel circulating miRNAs as biomarkers for Parkinson's disease | 3 years
  The study expects to discover novel circulating miRNAs as biomarkers for Parkinson's disease. As the deep phenotype characterization of the study sample, the project expects to identify new associations of identified miRNAs with disease-related parameters and define the role of miRNAs in the physiological pathways in which those parameters are involved and in the etiology of PD. Also, the understanding of the genetics of the disease will open avenues for novel therapeutic strategies

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ruggiero, Ph.D., Principal Investigator — Neuromed IRCCS
Locations (1):
- Neuromed IRCCS, Pozzilli, Molise, Italy